CLINICAL TRIAL: NCT03902847
Title: Efficacy of an Intensive Exercise Program Combined With Training on Action Observation and Motor Imagery for Improving Lumbopelvic Motor Control and Strengthening Trunk Muscles: A Randomized Controlled Trial
Brief Title: Motor Imagery and Action Observation on Lumbar Motor Variables
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 5
Record Dates: First submitted 2019-03-29; First posted 2019-04-04 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Motor Activity
Keywords: motor imagery; action observation; motor learning
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motor imagery (Experimental): All the subjects in this group were informed of the procedure at the beginning of the intervention, which consisted of the following: in the first phase (the first week), all participants had to perform the same motor control exercises program than the control group, but previously, a mental practice based on kinesthetic mental motor imagery was performed. To reinforce the process of motor imagery, a video with the exercises was shown to the subjects before performing the mental practice. All subjects had to imagine that he/she was performing each exercise during 1 set of 12 repetitions prior to the real execution of this. During the second phase (the second and third week), subjects had to complete the set both imagining, with visual mental motor imagery, and actively performing the exercises.
  Interventions: Behavioral: motor imagery
- Action observation (Experimental): All the subjects in this group were informed of the procedure at the beginning of the intervention, which consisted of the following: in the first phase (the first week), all participants had to perform the same motor control exercises program than the control group, but prior to the real execution, a video was shown in third-person perspective. All subjects watched one person performing each exercise during 1 set of 12 repetitions. During the second phase (the second and third week), subjects had to perform actively the exercises while they watched the video.
  All the participants also received a booklet with written information about the indications and exercises to be practiced at home to ensure that the training program was performed properly. Each week, participants received messages to remind and motivate them to undertake the exercise program daily.
  Interventions: Behavioral: Action observation
- Control group (Active Comparator): The subjects in this group received an intensive training program based on stabilization exercises of lumbo-pelvic region, which are common exercises used in rehabilitation of patients with chronic non-specific low back pain.
  Interventions: Behavioral: Motor Control Exercises

INTERVENTIONS:
Behavioral: motor imagery — All subjects had to imagine that he/she was performing each exercise during 1 set of 12 repetitions prior to the real execution of this. During the second phase (the second and third week), subjects had to complete the set both imagining, with visual mental motor imagery, and actively performing the exercises.
  Arms: Motor imagery
Behavioral: Action observation — A video was shown in third-person perspective. All subjects watched one person performing each exercise during 1 set of 12 repetitions. During the second phase (the second and third week), subjects had to perform actively the exercises while they watched the video.
  Arms: Action observation
Behavioral: Motor Control Exercises — The subjects were asked to perform 3 sets, of 10-12 repetitions each six exercise, with a total duration of approximately 30-35 minutes. The exercises program had to do it once a day, 6 days a week, for 3 weeks.
  Arms: Control group

SUMMARY:
Motor imagery is defined as a dynamic mental process of an action, without its real motor execution. Action observation evokes an internal, real-time motor simulation of the movements that the observer is perceiving visually. Both MI and AO have been shown to produce a neurophysiological activation of the brain areas related to the planning and execution of voluntary movement in a similar manner how the real action.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria were as follows:

* asymptomatic participants
* men and women aged 18 to 65 years.

Exclusion Criteria:

The exclusion criteria included the following:

* participants who had any knowledge of Physical Therapy or Occupational Therapy
* underage participants
* participants with any symptomatology in the lumbo-pelvic region at the time of the study -participants with lumbo-pelvic pain in at least the prior six months
* subjects who have been treated for lumbo-pelvic pain in the previous 6 months
* participants with any type of neurological disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Changes in the Right Lumbo-pelvic motor control | 1 week and 3 weeks
  Lumbar motor control will be measured by a pressure biofeedback called Stabilizer TM. The measurement protocol in the following procedure; The patient should be supine position with the Stabilizer TM placed in the lumbar region with an initial pressure of 70 mmHg. Then, the patient will be asked to flex the hip and knee at 90 ° with one leg and then with the opposite one. It is a validated and reliable protocol for motor control of the lumbar region
Changes in the Left Lumbo-pelvic motor control | 1 week and 3 weeks
  Lumbar motor control will be measured by a pressure biofeedback called Stabilizer TM. The measurement protocol in the following procedure; The patient should be supine position with the Stabilizer TM placed in the lumbar region with an initial pressure of 70 mmHg. Then, the patient will be asked to flex the hip and knee at 90 ° with one leg and then with the opposite one. It is a validated and reliable protocol for motor control of the lumbar region

SECONDARY OUTCOMES:
Perceived fatigue: changes in the Visual Analogue Scale-fatigue mid-intervention | 1 week and 3 weeks.
  Perceived fatigue will be measured with Visual Analogue Scale (VAS). The VAS consists of a 100-mm line, the left side of which represents "no fatigue" whereas the right side represents "maximal fatigue"
Changes in the trunk muscles strength | 1 week and 3 weeks.
  The strength of the lumbar region will be measured by a foot dynamometer (Takei TM 5420). The patient should stand on the dynamometer platform with knees extended, elbows extended, hips bent and index fingers holding the bar at knee height. Starting from this position the subject will have to make a previous adjustment of contraction of the musculature of the lumbar region and must perform a movement of lumbar extension. Subjects should maintain contraction for 3 seconds. It is a valid and reliable test to measure the muscular strength of the lumbar region

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No